CLINICAL TRIAL: NCT01412190
Title: An Open, Randomized, Single-centre, Intra-individual Controlled, Explorative, Safety and Efficacy Study Comparing Restylane Vital White With no Treatment in the Face, Back of the Hands and décolletage, Using an Injector Device
Brief Title: Study to Evaluate Restylane Vital Light Using an Injector Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31GR0803
Record Dates: First submitted 2011-06-30; First posted 2011-08-09 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2012-11

CONDITIONS: Aesthetics
Keywords: Skin rejuvenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Untreated (Other)
  Interventions: Other: No treatment
- Restylane Vital Light (Active Comparator): Restylane Vital Light administered at 3 treatment sessions 4 weeks apart
  Interventions: Device: Restylane Vital Light

INTERVENTIONS:
Device: Restylane Vital Light — Treatment of up to 4 ml for one side of the face, one hand and one side of the décolletage dispensed by 10ul doses 0.5-1 cm apart. 3 treatment sessions 4 weeks apart.
  Other Names: Restylane skinbooster
  Arms: Restylane Vital Light
Other: No treatment — One side of face, one hand and one side of the décolletage is left untreated as a control.
  Arms: Untreated

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of Restylane Vital White administered with an injector device on aged skin in the face, hands and décolletage.

DETAILED DESCRIPTION:
The objectives are to explore the safety and efficacy profile of Restylane Vital White administered with an injector device when one side of the face, one of the hands and one side of the décolletage is treated and the other side of the face, the other hand and the other side of the décolletage is left untreated. The face, the hands and the décolletage will be evaluated separately for both the efficacy and the safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained
* Female subjects 40-65 years of age, inclusive.
* Visible signs of skin aging in the face, hands and décolletage (e.g. reduced skin elasticity, reduced turgor, actinic elastosis, smaller and larger wrinkles) according to the Investigators opinion.
* Subjects must be cooperative and willing to comply with the instructions and procedures.

Exclusion Criteria:

* Extensively photo damaged and aged skin according to the Investigators opinion.
* Active skin disease, inflammation or related conditions, such as infection, perioral dermatitis, seborrheic eczema and rosacea in the face, hands or décolletage.
* History of or active collagenosis (e.g. systemic lupus, erythematosis, Rheumatic arthritis, skin or systemic sclerosis)
* Previous hypersensitivity to hyaluronic acid.
* Concomitant therapy with thrombolytics or anticoagulants, or have taken inhibitors of platelet aggregation, within 2 weeks before the baseline visit.
* History of cancerous or pre-cancerous lesions in the face, hands and décolletage.
* Previous tissue augmenting therapy with non-permanent filler or treatment with botulinum toxin, aesthetic surgical therapy, laser treatment, mesotherapy, or any form of peeling in the face, hands or décolletage within 12 months prior to the baseline visit.
* Use of injectable revitalization preparations (e.g. Hyal System®, Restylane Vital) within 12 months prior to the baseline visit.
* Use of retinoic acid within 6 months prior to the baseline visit.
* Previous or concomitant treatment with chemotherapy, immunosuppressive agents or corticoids.
* History of treatment with permanent filling materials.
* Pregnancy or breast feeding woman or woman of childbearing potential not practicing adequate contraception.
* Participation in any other clinical study within 30 days prior to the baseline visit or plan to participate in another clinical study during this study period.
* Unrealistic expectation with regard to the esthetic results of the treatment.
* Planned or ongoing weight reduction program during the study.
* Known history of drug or alcohol abuse within 6 months prior to the baseline visit.
* Known hypersensitivity to one or more components of EMLA cream®.
* Any medical condition that in the opinion of the Investigator makes the subject unsuitable for inclusion (e.g. severe chronic disease, malignancy, bleeding disorder, skin diseases etc).
* Other condition preventing the subject to entering the study in the Investigator's opinion e.g. subjects anticipated to be unreliable, unable to return for the follow-up visits, not likely to avoid other prohibited treatments or procedures or incapable of understanding the information or instructions.
* Nicotine use during the study or stopped within 12 months before the baseline visit.
* Study staff or close relative of study staff (e.g. parents, children, siblings and spouse).

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Elasticity | 0,4,8,12,20,28,36 weeks
  To evaluate the change in elasticity from baseline for the treated and untreated side respectively.
GEIS subject | 4,8,12,20,28,36 weeks
  To evaluate esthetic change from baseline as judged by the subjects using GEIS for the treated and untreated side respectively
GEIS blinded evaluator | 12,20,28,36 weeks
  To evaluate esthetic change from baseline as judged by the blinded evaluator using GEIS for the treated and untreated side respectively,
Skin structure | 0,4,8,12,20,28,36 weeks
  To evaluate the change in skin structure from baseline for the treated and untreated side respectively.
Subject satisfaction | 0,12,20,28,36 weeks
  To evaluate subject satisfaction
Best skin quality by blinded live evaluation | 12,20,28,36 weeks
  To evaluate best skin quality of treated and untreated side judged by a blinded live evaluation

SECONDARY OUTCOMES:
Adverse Events | 0-36 weeks
  To evaluate the safety of Restylane Vital White during the whole study by collecting Adverse Events
Subject diary | 2 weeks after each treatment
  To evaluate the acute safety profile, i.e. treatment procedure reactions by direct questioning to subjects in a diary used daily for 2 weeks after each injection.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Kerscher, Professor, Principal Investigator — University of Hamburg, Prof. Dr. Martina Kerscher, Department Chemie, Martin-Luther-King Platz 6, 20146 Hamburg
Locations (1):
- University of Hamburg, Hamburg, Germany